CLINICAL TRIAL: NCT00562497
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Prochymal® Infusion in Combination With Corticosteroids for the Treatment of Newly Diagnosed Acute GVHD
Brief Title: Efficacy and Safety of Prochymal® Infusion in Combination With Corticosteroids for the Treatment of Newly Diagnosed Acute Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 265
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Graft Versus Host Disease
Keywords: Acute GVHD; Acute Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — remestemcel-l; Adrenal Cortex Hormones; Methylprednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive 6 infusions of placebo-matching Prochymal® intravenously (IV) during the first 4 weeks of the study. The first infusion will be administered within 72 hours of the start of systemic corticosteroid therapy. Participants will receive 4 infusions during the first 2 weeks (twice weekly at least 3 days apart), followed by 2 infusions administered once weekly over the subsequent 2 weeks up to Day 28.
  Interventions: Other: Placebo; Other: Corticosteroid
- Prochymal® 2x10^6 hMSC/kg (Active Comparator): Participants will receive 6 infusions of Prochymal® 2x10^6 human mesenchymal stem cells (hMSC)/kg IV during the first 4 weeks of the study. The first infusion will be administered within 72 hours of the start of systemic corticosteroid therapy. Participants will receive 4 infusions during the first 2 weeks (twice weekly at least 3 days apart), followed by 2 infusions administered once weekly over the subsequent 2 weeks up to Day 28.
  Interventions: Drug: Prochymal®; Other: Corticosteroid

INTERVENTIONS:
Drug: Prochymal® — Prochymal® intravenous infusion.
  Other Names: Remestemcel-L
  Arms: Prochymal® 2x10^6 hMSC/kg
Other: Placebo — Placebo-matching Prochymal® intravenous infusion.
  Arms: Placebo
Other: Corticosteroid — Administration will be intravenously as prescribed by the caregiver.
  Other Names: Methylprednisolone; Prednisone

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled study to investigate the efficacy and safety of Prochymal® versus placebo in combination with corticosteroids as initial therapy for acute GVHD. Corticosteroids have been the primary therapy for patients with previously untreated acute GVHD and the historical published data define an expected 35% complete response (CR) at Day +28 using this therapy.

DETAILED DESCRIPTION:
Participants will be treated with a total of 6 infusions of investigational agent during the first 4 weeks of the study. The first infusion of the investigational product (IP) will be administered within 72 hours of the start of systemic corticosteroid therapy. Four infusions will be administered during the first two weeks (twice weekly), then two infusions administered during the next two weeks (once weekly). Participants assigned to the active treatment group will receive Prochymal®. Participants assigned to the non active treatment group will receive placebo (excipient, less cells). It is recommended that all participants receive all six infusions. The discontinuation of investigational agent is allowed for GVHD worsening with subsequent need for salvage therapy. All infusions must be given at least 3 days apart.

Participants will be evaluated for efficacy and safety until death, withdrawal or 90 study days after randomization, whichever occurs first. Study will be unblinded and data analyzed at Day 90 post 1st infusion (Day 0) following final participant enrollment. Participants will be followed for safety for 12 months post 1st infusion (Day 0).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years to 70 years of age, inclusive
* Participants must have received an allogeneic hematopoietic stem cell transplant using either bone marrow, peripheral blood stem cells or cord blood or administered a donor leukocyte infusion.
* Participants must have newly diagnosed Grades B-D acute GVHD. Biopsy confirmation of GVHD is strongly recommended but not required. Randomization should not be delayed awaiting biopsy or pathology results.
* Participants must be randomized and treated with corticosteroid (1-2 mg/kg/d methylprednisolone, or equivalent) and Prochymal®/placebo within 72 hours of onset of acute GVHD.
* Participants must have adequate renal function as defined by: Calculated Creatinine Clearance of >30 mL/min using the Cockcroft-Gault equation
* Participants who are women of childbearing potential, must be non-pregnant, not breast-feeding, and use adequate contraception. Male participants must use adequate contraception
* Participant must have a minimum Karnofsky Performance Level of at least 30 at the time of study entry
* Participant (or legal representative where appropriate) must be capable of providing written informed consent.

Exclusion Criteria:

* Participant has been previously treated with systemic immunosuppressive therapy for acute GVHD
* Participant has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant including uncontrolled infection, heart failure, pulmonary hypertension, etc.
* Participants may not receive any other investigational agents (not approved by the FDA for any indication) concurrently during study participation or within 30 days of randomization.
* Participant has a known allergy to bovine or porcine products or dimethyl sulfoxide (DMSO)
* Participant has received a transplant for a solid tumor disease.
* Participant requires more than 2 liters/min of oxygen to maintain stable oxygen saturation (Sa02) greater than or equal to 92%
* Participant requires a renal dopamine dose greater than 1-3 mcg/kg/min to maintain renal blood flow associated with renal failure and improved urinary output.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-01-31 (Actual); Primary Completion 2009-07-14 (Actual); Study Completion 2010-05-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Success | 90 Days
  Treatment was considered a success if all of the following conditions were met: Achieved induction of a complete response (CR) within 28 days after first infusion; CR followed by 28 days maintenance of a clinically meaningful response defined as the response that did not require an increase in corticosteroid dose (methylprednisolone doses >2 milligram/kilogram/day [mg/kg/d] or prednisone doses >2.5 mg/kg/d) for more than 7 consecutive days; Did not require second line/escalation therapy through Study Day 56; and survived 90 study days.

SECONDARY OUTCOMES:
Percentage of Participants with Overall Response | Day 90
  Overall Response was defined as participants who achieved complete response or partial response (CR+PR).
Percentage of Participants with Induction of a 2-grade decrease in (Graft Versus Host Disease) GVHD by Study Day 28 with maintenance of a 2-grade decrease in GVHD through Study Day 56 | Up to Day 56
Percentage of Participants with Induction of CR lasting for greater than or equal to 14 Days | Day 14
Percentage of Participants with Induction of a CR after Study Day 28 and clinically managed with steroids with second line/escalation therapy through Study Day 56 | Up to Day 56
Percentage of Participants with Induction of PR during the first 28 days | Up to Day 28
Time to achieve CR | Up to Day 90
Number of CR per organ | Up to Day 90
Total corticosteroid dose administered | Up to Day 90
Number of corticosteroid-related complications | Up to Day 90
  Corticosteroid-related complications included hyperglycemia requiring insulin, corticosteroid myopathy and psychosis.
Number of Infectious complications | Up to Day 90
  Infectious complications included viral, fungal or bacterial complications.
Number of Days of Hospitalization | Up to Day 90
Average Daily Corticosteroid Dose | Up to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Christopher James, PA, Study Director — Mesoblast, Inc.
Locations (53):
- United States (45):
  - University of Alabama Birmingham (UAB) Hospital, Birmingham, Alabama
  - UCLA Medical Center, Los Angeles, California
  - University of California Medical Center, San Francisco, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Hospitals, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Francis Cancer Center, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Medical Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Cancer Center, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Jewish Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center, University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Oncology Hematology Association, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Centers, Pittsburgh, Pennsylvania
  - Medical University of South Carolina(MUSC), Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - St. Vincent's Hospital, Darlinghurst
  - Royal Brisbane Hospital, Herston
- Canada (3):
  - Peter Lougheed Centre, Calgary, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- See also: Click here for more information about this study: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Prochymal® Infusion in Combination With Corticosteroids for the Treatment of Newly Diagnosed — http://www.osiris.com